CLINICAL TRIAL: NCT06414720
Title: Salivary MicroRNA in Endometriosis: Correlation With Progestin Treatment Response: A Prospective Observational Study
Brief Title: Salivary microRNA in Endometriosis: Correlation With Response to Progestin Therapy
Acronym: ENDOmiRNA
Status: Recruiting | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Giuseppe Vizzielli, Professor, University of Udine
Other Study IDs: ENDOmiRNA
Record Dates: First submitted 2024-05-05; First posted 2024-05-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; miRNA; Progesterone resistance
MeSH Terms: conditions — Endometriosis; Progesterone Resistance | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endometriosis patients: Patients diagnosed with endometriosis attending the Obstetrics and Gynecology Clinic at the Santa Maria della Misericordia Hospital in Udine, who have not yet started medical therapy.
  Interventions: Drug: Dienogest 2 MG

INTERVENTIONS:
Drug: Dienogest 2 MG — The patients will be started on progestin therapy after a saliva sample is collected from them for miRNA analysis.
  Other Names: zafrilla; devicius; endodien; visanne

SUMMARY:
This study aims to analyze the salivary miRNA specific for patients diagnosed with endometriosis, specifically evaluating the miRNA profile of patients who respond versus those who do not respond to progestin therapy. Ninety patients attending the Chronic Pelvic Pain Clinic will be recruited, and they will be asked to provide a saliva sample before starting medical therapy. The response to the therapy will be evaluated after 4 months from the beginning of the therapy itself.

DETAILED DESCRIPTION:
In recent years, scientific literature has focused on the search for new non-invasive diagnostic tools that can identify patients with endometriosis early and easily, thereby reducing diagnostic delay and enabling the immediate initiation of appropriate treatment. Among these, microRNA (miRNA) is emerging as a promising option. Despite recent progress in this field, a predictive biomarker of response to medical therapy or vice versa, resistance to progesterone in endometriosis, has not yet been identified, including among miRNAs. This study aims, therefore, to identify salivary miRNA signatures specific to endometriosis and differentially expressed between responder and non-responder patients to 2 mg dienogest medical therapy. 90 patients diagnosed with endometriosis attending the Obstetrics and Gynecology Clinic at the Santa Maria della Misericordia Hospital in Udine will be enrolled. The investigators will ask them for a salivary sample before starting the progestin therapy. After 4 months from the beginning, the response will be evaluated. The researchers will evaluate the differences between salivary miRNA of the responders vs non-responders.

ELIGIBILITY:
INCLUSION CRITERIA

* Age > 18 years
* Fertile age
* Clinical-ultrasound diagnosis or histological diagnosis of endometriosis
* Informed consent

EXCLUSION CRITERIA

* Pregnancy
* Pre-menarcheal or post-menopausal status
* Chronic pelvic pain syndrome with or without central sensitization assessed with the Central Sensitization Inventory Test (CSI)
* Neoplasia, diabetes, BMI > 30 kg/m2, coagulopathies, autoimmune diseases, or other conditions that may affect salivary miRNA measurement
* Currently undergoing progestin therapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients diagnosed with endometriosis attending the Obstetrics and Gynecology Clinic at the Santa Maria della Misericordia Hospital in Udine, who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
response to the progestin therapy | 0 (pre-therapy) - 4 months (after therapy)
  response to 2 mg dienogest therapy evaluated with NRS (numeric rating scale) scale assessed for acyclic pain, dyspareunia, dyschezia, dysmenorrhea, periovulatory pain
changes in quality of life | 0 (pre-therapy) - 4 months (after therapy)
  changes in quality of life assessed with questionnaire SF-36 (Short Form Health Survey 36)
differences in salivary miRNoma | sample collection at time 0, analysis after time 4
  Once it is established which patients are responders and which are non-responders, differential salivary miRNAs between the two groups will be identified via sequencing. The miRNA reverse transcription reaction will be performed using the reverse transcription kit TaqMan MicroRNA (Applied Biosystems). The reverse transcription product will be used for Real-time PCR. The small nucleolar RNA RNU6 will be used as an endogenous control. The protocol of Amplification will be carried out using the LightCycler 480 instrument (Roche). For each miRNA, qPCR will be performed in duplicate. The relative expression levels of miRNAs will be calculated using the 2-ΔΔCt method.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vizzielli, prof, Study Chair — University of Udine
Locations (1):
- University of Udine, Udine, UD, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bendifallah S, Suisse S, Puchar A, Delbos L, Poilblanc M, Descamps P, Golfier F, Jornea L, Bouteiller D, Touboul C, Dabi Y, Darai E. Salivary MicroRNA Signature for Diagnosis of Endometriosis. J Clin Med. 2022 Jan 26;11(3):612. doi: 10.3390/jcm11030612. PMID 35160066
- [Background] Zhang P, Wang G. Progesterone Resistance in Endometriosis: Current Evidence and Putative Mechanisms. Int J Mol Sci. 2023 Apr 10;24(8):6992. doi: 10.3390/ijms24086992. PMID 37108154
- [Background] Hon JX, Wahab NA, Karim AKA, Mokhtar NM, Mokhtar MH. MicroRNAs in Endometriosis: Insights into Inflammation and Progesterone Resistance. Int J Mol Sci. 2023 Oct 9;24(19):15001. doi: 10.3390/ijms241915001. PMID 37834449